CLINICAL TRIAL: NCT02031484
Title: Comparison of Continuous Sternal ECG Patch Monitors (Carnation and Zio) Trial
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Bardy Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Zio study
Record Dates: First submitted 2014-01-08; First posted 2014-01-09 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Syncope; Presyncope; Palpitations; Atrial Fibrillation; Supraventricular Tachycardia
MeSH Terms: conditions — Syncope; Atrial Fibrillation; Tachycardia, Supraventricular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is intended to compare the new Carnation patch monitoring system with the Zio patch, which represents the current standard for continuous recording of the ECG over extended periods.

DETAILED DESCRIPTION:
The purpose of this research is to confirm the clinical value of a new P-wave sensitive recording vector combined with an easy-to-use long-term cardiac rhythm monitoring patch system, the CarnationTM Ambulatory Monitoring (CAM) System. The P-wave is a critical aspect of the electrocardiogram and a key finding for proper arrhythmia diagnosis. The CAM system is optimized for both ease of use and for maximum P-wave clarity for arrhythmia diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Syncope of uncertain etiology or
* Pre-syncope of uncertain etiology or
* Palpitations of uncertain etiology or
* Management of known AF/SVT patients

Exclusion Criteria:

* Any dermatitis or infected skin over the sternum (Carnation patch) or left upper anterior thorax (Zio patch).
* A sternal or thoracic incision that extends under the patch within 3 months from the date of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in Chicago, Charlotte, and Iowa under the care of a physician for symptoms listed in the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-07; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
ECG signal quality | 14 days
  ECG signal quality = scoring the ability of each system to record electrical activity from the atrium (P-waves). The Physician Event Committee will independently score the P-waves from all recordings, using the following scale: Excellent, Good, Fair, Poor, Non-existent.

SECONDARY OUTCOMES:
Device comfort | 14 days
  Secondary outcome measures will include Human Factors performance of the 2 systems, which will be scored and compared in the following areas and duration of patch adherence: skin irritation, comfort, contact and stability.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kremers, MD, Principal Investigator — Mid Carolina Cardiology
Locations (4):
- United States (4):
  - University of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Mid Carolina Cardiology, Charlotte, North Carolina
  - Eastside Cardiology, Kirkland, Washington